CLINICAL TRIAL: NCT00085397
Title: A Randomized Phase II Study of Immunization Against Melanoma Comparing Autologous Dendritic Cells Pulsed With gp100 Peptide to Autologous Dendritic Cells Fused With Autologous Tumor Cells
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000369699; DFCI-03123
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2008-04

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma

ARMS (2):
- Arm I (Experimental): Patients undergo surgical harvesting of tumor cells for subsequent fusion. Patients receive vaccination comprising dendritic cells (DC) fused with autologous tumor cells subcutaneously on day 1. Treatment repeats every 21 days for 3 courses. Patients who achieve a partial (PR) or complete response (CR) may receive an additional 3 courses.
  Interventions: Biological: autologous dendritic cell-tumor fusion vaccine
- Arm II (Experimental): Patients receive vaccination comprising DC pulsed with gp100 antigen IV on day 1. Treatment repeats every 21 days for 6 courses. Patients who achieve a PR or CR may receive an additional 6 courses.
  Interventions: Biological: gp100 antigen; Biological: therapeutic autologous dendritic cells

INTERVENTIONS:
Biological: autologous dendritic cell-tumor fusion vaccine — Given subcutaneously
  Arms: Arm I
Biological: gp100 antigen — Given IV
  Arms: Arm II
Biological: therapeutic autologous dendritic cells — Given IV
  Arms: Arm II

SUMMARY:
RATIONALE: Vaccines made from a patient's dendritic cells may make the body build an immune response to kill tumor cells. It is not yet known whether combining vaccine therapy with either gp100 antigen or the patient's tumor cells will cause a stronger immune response and kill more tumor cells.

PURPOSE: This randomized phase II trial is studying vaccine therapy and gp100 antigen to see how well they work compared to vaccine therapy and patient's tumor cells in treating patients with stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the tumor-specific immune response, in terms of the number of gp100-specific cytotoxic T-lymphocytes, T-cell production of interferon gamma, or T-cell proliferation in response to in vitro exposure to gp100 and tumor lysate, in patients with stage III or IV melanoma treated with autologous dendritic cells (DC) pulsed with gp100 antigen vs autologous DC fused with autologous tumor cells.

Secondary

* Compare the safety and toxicity of these regimens in these patients.
* Compare the therapeutic effect of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

All patients undergo leukapheresis. Peripheral blood mononuclear cells are cultured to generate dendritic cells (DC).

* Arm I: Patients undergo surgical harvesting of tumor cells for subsequent fusion. Patients receive vaccination comprising DC fused with autologous tumor cells subcutaneously on day 1. Treatment repeats every 21 days for 3 courses. Patients who achieve a partial (PR) or complete response (CR) may receive an additional 3 courses.
* Arm II: Patients receive vaccination comprising DC pulsed with gp100 antigen IV on day 1. Treatment repeats every 21 days for 6 courses. Patients who achieve a PR or CR may receive an additional 6 courses.

In both arms, patients are followed monthly for 6 months.

PROJECTED ACCRUAL: A total of 40 patients (20 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous melanoma

  * Stage III or IV disease
  * Recurrent or de novo stage III disease allowed if disease is unresectable and no definitive treatment is available
* gp100- and HLA-A201-positive
* Surgically accessible tumor, defined by 1 of the following:

  * Pulmonary lesions approachable by thoracoscopic procedure
  * Skin or superficial soft tissue or lymph node lesions amenable to resection under local anesthesia
  * Malignant ascites or pleural effusion
* Measurable disease in addition to surgically accessible tumor > 2.0 cm
* No CNS metastases
* No mucosal or ocular melanoma

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* WBC > 3,000/mm^3
* Platelet count > 75,000/mm^3

Hepatic

* Bilirubin < 2.0 mg/dL

Renal

* Creatinine < 2.0 mg/dL

Immunologic

* No active infection requiring treatment
* No clinically significant autoimmune disorder
* No immune deficiency disorder
* HIV negative

Other

* Antecubital vein accessible for leukapheresis
* No other malignancy within the past 5 years except nonmelanoma skin cancer or squamous cell carcinoma in situ of the cervix
* No pre-existing comorbid disease that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior melanoma vaccine therapy
* More than 6 weeks since prior immunotherapy

Chemotherapy

* No prior chemotherapy for metastatic melanoma

Endocrine therapy

* No concurrent corticosteroids

Radiotherapy

* More than 6 weeks since prior radiotherapy

Surgery

* Not specified

Other

* No concurrent systemic immunosuppressive therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-03

PRIMARY OUTCOMES:
Immune response

CONTACTS AND LOCATIONS:
Overall Officials: Frank Haluska, MD, PhD, Principal Investigator — Massachusetts General Hospital; David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts